CLINICAL TRIAL: NCT05549492
Title: Transversus Abdominis Plane Block With or Without Buprenorphine After Inguinal Hernia Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nirvana Ahmed 01
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Inguinal Hernia; Pain, Postoperative
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Ropivacaine; Buprenorphine

STUDY DESIGN:
Intervention Model Description: to determine if TAP block treatment, either with or without buprenorphine, affected patients having inguinal hernias repaired
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (Experimental): Candidates received 20 ml of 0.25% ropivacaine for TAP block
  Interventions: Drug: Ropivacaine 0.25%-NaCl 0.9% Injectable Solution
- Group RB (Experimental): Candidates received 20 ml of 0.25% ropivacaine and 300 μg of buprenorphine, respectively, for the TAP block.
  Interventions: Drug: Ropivacaine 0.25%-NaCl 0.9% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.25%-NaCl 0.9% Injectable Solution — The pain level of the cases is evaluated by means of the digital pain (numeric rating) scale from 0 to 10 in which 0 means "no pain" and 10 means "the worst pain" as well as the duration of pain relief and the need for another dose of the same analgesic or other. The pain level is evaluated again if it is present.
  Other Names: buprenorphine 300 μg

SUMMARY:
Buprenorphine intravenous, sublingual, and transdermal patches have been researched for their antihyperalgesic effects, although peripherally mediated effects have not been examined in Egypt surprisingly

DETAILED DESCRIPTION:
This prospective, randomized, double-blind controlled trial involved 88 patients who were scheduled for inguinal hernia surgery followed by a TAP block. Patients were allocated into group B (n= 44) received 20 ml of 0.25% Ropivacaine for TAP block; group BR (n= 44) received 20 ml of 0.25% Ropivacaine containing 300 μg of buprenorphine for TAP Block. The primary outcome of the study was the analgesic and antihyperalgesic effect of buprenorphine compared to the control group. The duration of analgesia, analgesic consumption, postoperative pain scores at rest and sitting up to 48 hrs, and effect on wound hyperalgesia at 24 and 48 hrs were evaluated. Secondary outcomes of the study include incidence of side effects and TAP block-related complications were recorded. Effect of buprenorphine on patients with predicted high pain scores and incidence of persistent postoperative pain were also determined.

A transversus abdominis plane (TAP) block provides analgesia of the anterior and lateral abdominal wall below the umbilicus by blocking the T6-L1 segmental nerves as they lie within the fascial plane between the transversus abdominis and internal oblique muscles: bilateral block for midline abdominal incision. It was first described in 2001 by Rafi as a traditional blind landmark technique using the lumbar triangle of Petit. Local anesthetic is then injected between the internal oblique and transverse abdominis muscles just deep the fascial plane, the plane through which the sensory nerves pass

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Inguinal Hernia
2. Medically free

Exclusion Criteria:

1. participants with a history of heart, renal and liver cell failure.
2. allergic reaction to studied drugs, and history of epilepsy,
3. hydrodynamic instability,
4. chronic pain.
5. mental illness.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Post Operative Pain | 2 hours after the operation upto 48-hour analgesic after surgery
  The pain level of the cases is evaluated by means of the digital pain as the 11-point visual analog scale (VAS) whereas 0-Represents no pain, 10 - Worst imaginable pain), as well as the 11-point VAS-A (0-Represents no anxiety, 10 - Highest anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Nirvana Elshalakany, Professor, Principal Investigator — Department of Anesthesia and I.C.U. faculty of Medicine October six university, Egypt
Locations (1):
- October 6 University Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided